CLINICAL TRIAL: NCT03969381
Title: Diffusion-weighted Magnetic Resonance Imaging in Post Therapy Evaluation of Patients With Malignant Lymphoma: Comparison With 2-deoxy-2-fluoro-D-glucose-positron Emission Tomography/Computed Tomography
Brief Title: Diffusion-weighted Magnetic Resonance Imaging in Post Therapy Patients With Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Ali Gamal, principel investigator, Assiut University
Other Study IDs: lymphoma
Record Dates: First submitted 2019-05-23; First posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1 lymphoma patients: pre therapy and post therapy of lymphoma patients
  Interventions: Radiation: diffusion weighted magnetic resonance image in lymphoma

INTERVENTIONS:
Radiation: diffusion weighted magnetic resonance image in lymphoma — compare between result of positron emission tomography /computed tomography and diffusion weighted imaging in followup of lymphoma

SUMMARY:
* The goal of this study is to determine the feasibility of the diffusion weighted Magnetic Resonance Imaging in the evaluation of the treatment response in patients with malignant lymphoma.
* The investigator's objective is to compare the changes of mean Apparent Diffusion Coefficient value of the tumor with the changes of maximum Standardized Uptake Value of the tumor in positron Emission Tomography Computed Tomography in both pre and post therapy status .

DETAILED DESCRIPTION:
Lymphomas are the malignant tumors of lymph nodes and considered as one of the most common primary hematopoietic malignancy. Multi slice computed tomography is the most readily available and most commonly used tool for staging lymphoma. But it has multiple limitations in diagnosis of lymphoma as the recognition of lymph node involvement is based only on the size of the lymph node without any metabolic information .

The tumors rely on glucose as their substrate for energy production and replication, this metabolic information can be obtained from the 2-deoxy-2-fluoro-D-glucose Among the positron Emission Tomography Computed Tomography parameters, standardized uptake value is currently the most commonly used semi-quantitative index of 2-deoxy-2-fluoro-D-glucose metabolic rate. standardized uptake value reflects tumor glucose metabolism, and is commonly represented by the maximum standardized uptake value .2-deoxy-2-fluoro-D-glucose positron Emission Tomography Computed Tomography has been shown to be more accurate for the evaluation of the extent of disease and treatment response by providing these metabolic information in patients with malignant lymphoma .

2-deoxy-2-fluoro-D-glucose positron Emission Tomography Computed Tomography , with the advantage of being able to perform whole-body detection of malignant lesions, is considered to be the current standard of practice for the management of lymphomas; however, positron Emission Tomography Computed Tomography is expensive, time-consuming, involves exposure to ionizing radiation and is not widely available because it requires large and expensive equipment . In contrast, Magnetic Resonance Imaging provides excellent tissue contrast, high spatial resolution, detailed morphological information without the use of ionizing radiation . Diffusion-weighted Magnetic Resonance Imaging is a noninvasive technique allows visualization of diffusion properties of water molecules in biologic tissues. .

A supplemental tool in Diffusion-weighted imaging is the apparent diffusion coefficient map , acquired by post-processing of the obtained Diffusion-weighted images . apparent diffusion coefficient allows for quantitative definition of diffusion parameters (in mm2/sec) . Diffusion-weighted images with apparent diffusion coefficient mapping could provide useful functional information regarding the characterization of lymphomas .Because of their high cellularity and high nuclear-to-cytoplasm ratio .

ELIGIBILITY:
Inclusion Criteria:

* patients clinically diagnosed as lymphoma patient can tolerate the magnetic resonance examination.

Exclusion Criteria:

* presence of paramagnetic substance as peace maker or cochlear implants and claustrophobia.

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed as malignant lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
role of diffusion weighted imaging in followup of lymphoma | 5 minutes
  • measures mean Apparent diffusion coefficient value in pre and post therapy status in patients with lymphoma with cut off value 1 .

CONTACTS AND LOCATIONS:
Overall Officials: sara, Msc, Principal Investigator — Assiut University